CLINICAL TRIAL: NCT03645564
Title: Impact of the Information Follow-up Given to Patients on Their Disease Understanding and Therapeutic Adherence in Patients Under Direct Oral Anticoagulants and With Atrial Fibrillation in a Cardiology Department
Acronym: RYTHM-UP AOD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment incomplete due to COVID
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2016/43
Record Dates: First submitted 2018-08-20; First posted 2018-08-24 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation
Keywords: Stroke; Anti-vitamin K; Direct anti-coagulant; Nurse
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Intervention Model Description: It is an open, prospective, randomized, 2 arms study that will compare 2 groups of patients care for Atrial Fibrillation in the Cardiology-Electrophysiology and Cardiac Stimulation Department with direct oral anticoagulants prescription.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : specialized nurse consultation (Active Comparator): This group will benefit of a specialized nurse consultation throughout of which an individualized information will be delivered. This information will be reevaluated during the usual patient follow-up.
  Interventions: Other: Specialized nurse consultation
- Group 2 : no specialized nurse consultation (No Intervention): This control group will present the same care pathway than all the patients of the service suffering from Atrial Fibrillation without specialized nurse consultation.

INTERVENTIONS:
Other: Specialized nurse consultation — The purpose of this consultation is to establish a partnership between the patient and the nursing staff. Tools were set up (notebook, movie) to answer the questions of the patient. In case of specific question, an expert will meet the patient (doctor of the service, psychologist, pharmacist or hematologist).
  Arms: Group 1 : specialized nurse consultation

SUMMARY:
The primary objective of this study is to measure in patients addressed for Atrial Fibrillation (AF) in the Cardiology-Electrophysiology and Cardiac Stimulation Department of Bordeaux hospital, the impact of a specialized nurse consultation on their adherence level to direct oral anticoagulants treatments.

DETAILED DESCRIPTION:
The number of persons that should take an anticoagulant treatment in France is evaluated at 3 Billion and at least half of them for an Atrial Fibrillation disease. One of the main issues of their prescription is stoke prevention. With the coming of direct oral anticoagulants, which does not require repeating controls like it is the case for anti-vitamin K treatments, the patient's involvement is a guarantee of therapeutic adherence and good use. Nevertheless a good adherence level is seldom reached. This highlights the importance of individualized information which must be followed for purposes of accuracy and deepening. Thus as part of investigator's activity department that treats about 1000 patients per year for an Atrial Fibrillation, the information, use and therapeutic adherence are a priority in the care pathway of patients under direct oral anticoagulants. The investigators propose to measure the contribution of a specialized nurse consultation in contact with a multidisciplinary team on therapeutic adherence. The investigators hypothesis that an individualized and reassessed information would allowed a better understanding by the patients of their pathology and care and thus a better therapeutic adherence. A control group will present the same care pathway than all the patients of the service suffering from Atrial Fibrillation without specialized nurse consultation. The second group will benefit of a specialized nurse consultation throughout of which an individualized information will be delivered. This information will be reevaluated during the usual patient follow-up. All the patients will be followed at 3 months, 6 months and 1 year as part of the usual care of the service.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in the Cardiology-Electrophysiology and Cardiac Stimulation Department for an AF,
* Patient requiring direct oral anticoagulant treatment,
* Age ≥ 18 years of both genders,
* Written consent,
* Patient affiliated or beneficiary of a social insurance,
* French language.

Exclusion Criteria:

* Patient unable to give his written consent or with cognitive disorders,
* Patient depending of a third person,
* Patient unable to be followed in the service,
* Patient in exclusion period for another protocol,
* Subject deprived of liberty by judicial or administrative decision,
* Protected adults,
* Non-inclusion criteria specific to direct oral anticoagulants (valvular AF, severe renal impairment).

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Adherence to direct oral anticoagulants | 12 months
  Adherence questionnaire

SECONDARY OUTCOMES:
Change in the level of knowledge of disease and treatment | Change from baseline at 12 months
  Assessment by auto-questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie PETIT-MONEGER, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Pessac, France